CLINICAL TRIAL: NCT01396044
Title: Daily Checklists and Outcome in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Parker B. Francis Fellowship Program (Unknown)
Responsible Party: Principal Investigator, Curtis Weiss, Instructor of Medicine, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NUIRBSTU00013313
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Critical Illness
Keywords: Quality improvement; Checklist; Critical care; Anti-bacterial agents; Mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic checklist (Experimental): Electronic checklist
  Interventions: Other: Electronic checklist
- Verbal prompting (Experimental): Verbal prompting with written checklist
  Interventions: Other: Verbal prompting

INTERVENTIONS:
Other: Electronic checklist — Electronic checklist for process of care issues implemented in our institution. Training on a regular basis of the electronic checklist arm to use the electronic checklist. Process of care issues on the electronic checklist include several that are under investigation: antibiotics and mechanical ventilation.
  Arms: Electronic checklist
Other: Verbal prompting — Prompting by study investigators of physicians on the verbal prompting arm. Prompting will include questions related to antibiotic utilization and mechanical ventilation weaning.
  Arms: Verbal prompting

SUMMARY:
Medical errors account for tens of thousands of deaths and tens of billions of dollars in healthcare costs in the United States every year. One field that has seen the strongest push toward quality improvement has been critical care medicine, likely because its particularly high degree of medical complexity makes it a practice area prone to high error rates with serious consequences. One of the most commonly used interventions used to help reduce errors in the intensive care unit (ICU) has been the implementation of checklists.

The investigators propose a clinical trial in a University critical care setting to determine whether an electronic checklist versus verbal prompting to use a written checklist improves clinical practice and patient outcomes. The investigators also plan to compare these data with a time period prior to the study to determine if the electronic checklist or verbal prompting are better than usual care. The investigators hypothesize that both the electronic checklist and verbal prompting to use a written checklist will be better for clinical practice and patient outcomes than usual care, and that verbal prompting will lead to better outcomes compared to the electronic checklist.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a medical intensive care unit (MICU) team during the study timeframe

Exclusion Criteria:

* Transfer from MICU team to a separate ICU team within 12 hours of admission
* Transfer to MICU team from a separate ICU team after more than 72 hours on the separate ICU team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis H Weiss, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

REFERENCES:
- [Background] Weiss CH, Moazed F, McEvoy CA, Singer BD, Szleifer I, Amaral LA, Kwasny M, Watts CM, Persell SD, Baker DW, Sznajder JI, Wunderink RG. Prompting physicians to address a daily checklist and process of care and clinical outcomes: a single-site study. Am J Respir Crit Care Med. 2011 Sep 15;184(6):680-6. doi: 10.1164/rccm.201101-0037OC. Epub 2011 May 26. PMID 21616996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients admitted to the MICU service at Northwestern Memorial Hospital on or after June 27, 2011 and discharged on or prior to October 7, 2011 were enrolled. Exclusion criteria: patients transferred to or from a different ICU service, and MICU re-admission without intervening hospital discharge.
Pre-assignment Details: Patients were included only if they were treated with at least one day of empirical antibiotics.
Period: Overall Study
Arm/Group | Electronic Checklist | Verbal Prompting
Started | 125 | 171
Completed | 125 | 171
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electronic Checklist | Verbal Prompting | Total
Number analyzed (Participants) | 125 | 171 | 296
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 101 | 165
  >=65 years | 61 | 70 | 131
Age Continuous [Mean (Standard Deviation); unit: years] | 62.6 (17.6) | 60.0 (17.8) | 61.1 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 83 | 142
  Male | 66 | 88 | 154
Region of Enrollment [Number; unit: participants]
  United States | 125 | 171 | 296

OUTCOME MEASURES:

1. Primary Outcome: Empiric Antibiotic Duration
Time Frame: During intensive care unit admission, an average of 5 days per patient (although individual patients may vary)
Population: All patients who received at least one day of empirical antibiotics during their ICU admission.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
days | 3 [2 to 4] | 3 [1 to 5]
Statistical Analysis 1: Comparison: Electronic Checklist vs Verbal Prompting; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Proportion of Empiric Antibiotics
Description: The difference between the electronic checklist and prompted groups' proportion of all antibiotics that were administered empirically (empiric/total antibiotics).
Time Frame: ICU admission
Population: All patients who received at least one day of empirical antibiotics during their ICU admission.
Measure: Mean (Standard Deviation); unit: proportion of antibiotic-days
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
proportion of antibiotic-days | 0.83 (0.27) | 0.78 (0.27)
Statistical Analysis 1: Comparison: Electronic Checklist vs Verbal Prompting; Test type: Superiority or Other; p = 0.093, t-test, 2 sided

3. Secondary Outcome: Hospital Mortality
Time Frame: During hospitalization, an average of 2 weeks per patient (although individual patients may vary)
Population: All patients treated with at least one day of empirican antibiotics during ICU admission
Measure: Number; unit: number of deaths
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
number of deaths | 30 | 30
Statistical Analysis 1: Comparison: Electronic Checklist vs Verbal Prompting; Test type: Superiority or Other; p = 0.17, Chi-squared

4. Secondary Outcome: Length of Stay
Time Frame: During hospitalization, an average of 2 weeks per patient (although individual patients may vary)
Population: All patients treated with at least one day of empirical antibiotics.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
days | 2.8 [1.7 to 6.5] | 2.6 [1.5 to 6.9]
Statistical Analysis 1: Comparison: Electronic Checklist vs Verbal Prompting; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Ventilator-free Days
Description: Number of days within the first 28 days after ICU admission that a patient does not require mechanical ventilation.
Time Frame: During hospitalization, an average of 2 weeks per patient (although individual patients may vary)
Population: All patients treated with at least one day of empirical antibiotics.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
days | 20.3 [0 to 25.9] | 21.9 [13.5 to 25.7]
Statistical Analysis 1: Comparison: Electronic Checklist vs Verbal Prompting; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Proportion of Successful Prompts
Description: Prompting group: number of patient-days that prompting led to empirical antibiotics being discontinued or narrowed/number of patient-days prompting occurred
  Electronic checklist group: number of patient-days that electronic checklist led to empirical antibiotics being discontinued or narrowed/number of patient-days electronic checklist was completed
Time Frame: During ICU admission, an average of 5 days (although individual patients may vary)
Population: All patients treated with at least one day of empirical antibiotics.
Measure: Number; unit: proportion of patient-days
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
proportion of patient-days | 0.096 | 0.436

7. Secondary Outcome: Proportion of Patients-days on Which Empirical Antibiotics Were Used
Description: Proportion of patients-days on which empirical antibiotics were used
Time Frame: ICU admission
Population: All patients who received at least one day of empirical antibiotics.
Measure: Number; unit: Number of patient-days
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
Number of patient-days | 498 | 702
Statistical Analysis 1: Comparison: Electronic Checklist vs Verbal Prompting; Test type: Superiority or Other; p = 0.002, Chi-squared

8. Secondary Outcome: Standardized Mortality Ratio
Time Frame: Hospital admission
Population: All patients treated with at least one day of empirical antibiotics.
Measure: Mean (95% Confidence Interval); unit: observed/expected deaths
Arm/Group | Electronic Checklist | Verbal Prompting
Number analyzed (Participants) | 125 | 171
observed/expected deaths | 0.70 [0.47 to 1.0] | 0.64 [0.43 to 0.92]

ADVERSE EVENTS:
Arm/Group | Electronic Checklist | Verbal Prompting
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/171
Other Adverse Events (participants affected / at risk) | 0/125 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No